CLINICAL TRIAL: NCT02684474
Title: Expanded Access Protocol Using HBOC-201 to Treat Patients With Life Threatening Anemia, for Whom Blood is Not an Option
Brief Title: Expanded Access Protocol Using HBOC-201
Status: No longer available | Type: Expanded Access
Sponsor: Johns Hopkins University (Other)
Collaborators: HbO2 Therapeutics LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: IRB00090805
Record Dates: First submitted 2016-02-10; First posted 2016-02-18 (Estimated); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — HBOC 201

INTERVENTIONS:
Biological: HBOC-201 — Intravenous administration of a hemoglobin based oxygen carrier (HBOC) in patients with life-threatening anemia, for whom allogeneic blood transfusion is not an option.
  Other Names: Hemopure

SUMMARY:
The purpose of this protocol is to provide treatment with HBOC-201 to patients with life-threatening anemia for whom allogeneic blood transfusion is not an option. HBOC 201 [hemoglobin glutamer - 250 (bovine)] has been previously studied as an alternative to blood transfusions in severely anemic patients needing a way to enhance tissue oxygenation. HBOC-201 is purified, cross-linked and polymerized acellular bovine hemoglobin in a modified lactated Ringer's solution, and does not require blood compatibility.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 18 years of age
2. Critically ill patients with hemoglobin ≤ 6 g/dL (or 7-8 g/dL with significant active bleeding), and physiologic evidence of critical ischemia, for example: elevated troponins, altered mental status, acute renal failure, lactic acidosis or evidence of central nervous system acute deficits
3. Patients or their Legally Authorized Representative who are able and willing to provide informed consent
4. Blood is not an option due to:

   * refusal of transfusion
   * lack of compatible red blood cells

Exclusion Criteria:

1. Patients with known hypersensitivity or allergy to beef products
2. Patients with pre-existing uncontrolled hypertension, heart failure, renal failure, circulatory hypervolemia or systemic mastocytosis*
3. Patients who are eligible for blood transfusions
4. Patients who are > 80 years old*

   * on a case by case and quality of life determination

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Steven M Frank, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- The Johns Hopkins Hospital, Baltimore, Maryland, United States

REFERENCES:
- [Background] Frank SM, Wick EC, Dezern AE, Ness PM, Wasey JO, Pippa AC, Dackiw E, Resar LM. Risk-adjusted clinical outcomes in patients enrolled in a bloodless program. Transfusion. 2014 Oct;54(10 Pt 2):2668-77. doi: 10.1111/trf.12752. Epub 2014 Jun 18. PMID 24942198
- [Background] Resar LM, Frank SM. Bloodless medicine: what to do when you can't transfuse. Hematology Am Soc Hematol Educ Program. 2014 Dec 5;2014(1):553-8. doi: 10.1182/asheducation-2014.1.553. Epub 2014 Nov 18. PMID 25696910
- [Background] Chaturvedi S, Koo M, Dackiw L, Koo G, Frank SM, Resar LMS. Preoperative treatment of anemia and outcomes in surgical Jehovah's Witness patients. Am J Hematol. 2019 Feb;94(2):E55-E58. doi: 10.1002/ajh.25359. Epub 2018 Dec 18. No abstract available. PMID 30474135
- [Background] Resar LM, Wick EC, Almasri TN, Dackiw EA, Ness PM, Frank SM. Bloodless medicine: current strategies and emerging treatment paradigms. Transfusion. 2016 Oct;56(10):2637-2647. doi: 10.1111/trf.13736. Epub 2016 Jul 29. PMID 27473810
- [Background] Visagie M, Pearson KR, Purvis TE, Gehrie EA, Resar LMS, Frank SM. Greater anemia tolerance among hospitalized females compared to males. Transfusion. 2019 Aug;59(8):2551-2558. doi: 10.1111/trf.15338. Epub 2019 May 7. PMID 31063596
- [Background] Frank SM, Chaturvedi S, Goel R, Resar LMS. Approaches to Bloodless Surgery for Oncology Patients. Hematol Oncol Clin North Am. 2019 Oct;33(5):857-871. doi: 10.1016/j.hoc.2019.05.009. Epub 2019 Jul 31. PMID 31466609
- [Background] Guinn NR, Resar LMS, Frank SM. Perioperative Management of Patients for Whom Transfusion Is Not an Option. Anesthesiology. 2021 Jun 1;134(6):939-948. doi: 10.1097/ALN.0000000000003763. No abstract available. PMID 33857295
- [Background] Frank SM, Pippa A, Sherd I, Scott AV, Lo BD, Cruz NC, Hendricks EA, Ness PM, Chaturvedi S, Resar LMS. Methods of Bloodless Care, Clinical Outcomes, and Costs for Adult Patients Who Decline Allogeneic Transfusions. Anesth Analg. 2022 Sep 1;135(3):576-585. doi: 10.1213/ANE.0000000000006114. Epub 2022 Aug 17. PMID 35977366
- [Background] Cruz NC, Guinn NR, Adegboye J, Hsiao J, Thomas AJ, Lo BD, Chaturvedi S, Resar LMS, Frank SM. A novel algorithm to calculate target preoperative hemoglobin for patients declining allogeneic transfusion. J Clin Anesth. 2023 Aug;87:111070. doi: 10.1016/j.jclinane.2023.111070. Epub 2023 Feb 27. No abstract available. PMID 36857836
- [Background] Asiedu JO, Thomas AJ, Cruz NC, Nicholson R, Resar LMS, Khashab M, Frank SM. Management and clinical outcomes for patients with gastrointestinal bleeding who decline transfusion. PLoS One. 2023 Aug 25;18(8):e0290351. doi: 10.1371/journal.pone.0290351. eCollection 2023. PMID 37624779
- [Background] Sklar MB, Kajstura TJ, Vogt SL, Gray C, Ulatowski JA, Resar LMS, Frank SM. Gastrointestinal Bleeding and Survival After a Nadir Hemoglobin <3.0 g/dL in 2 Jehovah's Witness Patients: A Case Report. A A Pract. 2024 Aug 13;18(8):e01837. doi: 10.1213/XAA.0000000000001837. eCollection 2024 Aug 1. PMID 39137122
- [Background] Lo BD, Pippa A, Sherd I, Scott AV, Thomas AJ, Hendricks EA, Ness PM, Chaturvedi S, Resar LMS, Frank SM. Clinical Outcomes, Blood Utilization, and Ethical Considerations for Pediatric Patients in a Bloodless Medicine and Surgery Program. Anesth Analg. 2024 Feb 1;138(2):465-474. doi: 10.1213/ANE.0000000000006776. Epub 2024 Jan 12. PMID 38175737